CLINICAL TRIAL: NCT00693940
Title: Increasing Activity in Peripheral Arterial Disease
Brief Title: Effectiveness of Group Walking Sessions for Increasing Activity in People With Peripheral Arterial Disease (The Group Oriented Arterial Leg Study [GOALS])
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary McDermott, Professor of Medicine and Preventive Medicine at Northwestern University Feinberg School of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 586; R01HL088589-01 (NIH); HL088589-01
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Peripheral Vascular Diseases; Cardiovascular Diseases
Keywords: Peripheral Arterial Disease; PAD
MeSH Terms: conditions — Peripheral Vascular Diseases; Cardiovascular Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive treatment with group mediated cognitive behavioral sessions.
  Interventions: Behavioral: Group mediated cognitive behavioral (GMCB) sessions
- 2 (Active Comparator): Participants will receive treatment with health education sessions.
  Interventions: Other: Health education sessions

INTERVENTIONS:
Behavioral: Group mediated cognitive behavioral (GMCB) sessions — GMCB will include weekly group exercise sessions, lasting approximately 60 to 75 minutes each for a 6 month period. During these sessions, participants will be asked to exercise by walking around a track. There will also be a group discussion, led by a facilitator, who will help participants find ways to increase the frequency of their walking exercise at home. After completing the GMCB sessions, which will last about 6 months, participants will be telephoned regularly by a study coordinator for another 6 months.
  Arms: 1
Other: Health education sessions — Health education will include weekly educational sessions on a health-related topic, lasting approximately 60 minutes each. After completing the health education sessions, which will last about 6 months, participants will be telephoned regularly by a study coordinator for another 6 months.
  Arms: 2

SUMMARY:
Lower extremity peripheral arterial disease (PAD) is a disease in which fatty build-up, or plaque, accumulates in the arteries of the legs. People with lower extremity PAD often experience leg pain while walking, which is caused by reduced blood flow to the legs. Regular walking has significant benefits for people with blood flow problems in their legs, but previous studies have shown that most men and women with PAD do not walk for exercise on a regular basis. A group home-based walking program may help people with PAD to walk more often and improve their lower extremity functioning. This study will evaluate the effectiveness of a home-based group mediated cognitive behavioral (GMCB) exercise program in helping people with lower extremity PAD to increase their walking frequency and improve their lower leg functioning.

DETAILED DESCRIPTION:
Lower extremity PAD affects between 10% and 15% of people over the age of 65. A person's risk for PAD increases with age but can also be raised by smoking or having diabetes, high blood pressure, high cholesterol, or heart disease. PAD symptoms may include leg pain, foot or toe wounds, and a noticeably lower temperature in the lower legs than in the rest of the body. The specific functional impairments caused by PAD symptoms are associated with increased risks of disability, nursing home placement, mobility loss, hospitalization, and mortality. Supervised exercise rehabilitation programs have been shown to improve walking ability in people with PAD. However, few people with PAD have access to supervised exercise rehabilitation programs because of costs and difficulty traveling to the exercise facility. Home-based exercise programs may be more beneficial than supervised programs in improving lower extremity functioning in people with PAD, but more information is needed to support the effectiveness of at-home rehabilitation. This study will compare the effectiveness of a home-based GMCB exercise program versus general health education sessions in helping people with lower extremity PAD to increase their walking frequency and improve their lower leg functioning.

Participation in this study will last 12 months. The primary outcome will be measured at 6 month follow-up. All participants will undergo a baseline 6-minute walk test on a treadmill and an electrocardiogram (ECG). They will also provide information on their physical activity levels. Participants will then be assigned randomly to receive GMCB sessions or health education sessions. Both groups will attend weekly sessions of their assigned treatment for a 6 month period. During the GMCB sessions, participants will be asked to exercise by walking around a track. There will also be a group discussion, led by a facilitator, who will help participants find ways to increase the frequency of their walking exercise at home. Each GMCB session will last approximately 60 to 75 minutes. Health education sessions will last 60 minutes and will cover health-related topics.

After completing approximately 6 months of treatment, participants in both groups will be telephoned regularly by a study coordinator: they will receive telephone calls every other week during Months 6 to 9 of follow-up and monthly during Months 9 to 12 of follow-up. Participants will be asked to return for follow-up testing at Month 6 and Month 12; outcomes measured at Month 6 are highest priority.

ELIGIBILITY:
Inclusion Criteria:

* Have PAD
* Potential participants with a resting ABI greater than or equal to 0.91 and less than or equal to 1.00 at their baseline visit will be eligible if their ABI drops by at least 20% after the heel-rise test. Potential participants with a resting baseline ABI greater than 0.91 who do not meet criteria for inclusion based on the heel-rise test can be eligible if they have data from a certified non-invasive vascular laboratory that demonstrates presence of lower extremity ischemia. However, more evidence than an abnormal PVR from the non-invasive vascular laboratory is required (for example, a toe brachial index pressure less than 0.60). Finally, potential participants who do not meet the above criteria for inclusion will be eligible if they have an angiogram demonstrating greater than 50% stenosis on one or more lower extremity arterial vessels.

Exclusion Criteria:

* Below or above knee amputation
* Wheelchair confinement
* Uses a walking aid other than a cane (e.g., walker)
* Unable to return to the medical center at the required visit frequency
* Greater than Class II New York Heart Association heart failure or angina (symptoms at rest or with minimal exertion)
* Any increase in angina pectoris symptoms during the 6 months before study entry or angina at rest
* Presence of a foot ulcer
* Lower extremity revascularization or major orthopedic surgery during the 3 months before study entry
* Heart attack or coronary artery bypass grafting during the 3 months before study entry
* Major medical illnesses, including treatment for cancer (except non-melanoma skin cancer) during the 12 months before study entry
* Planned lower extremity revascularization within the 12 months after study entry
* Current participation in another clinical trial
* Walking for exercise at a level comparable to that targeted in the study's intervention
* Completion of a cardiac rehabilitation program within 3 months before study entry
* Coronary ischemia during exercise, defined as ST segment depression greater than 1 mm during the baseline exercise treadmill test, with or without associated chest discomfort
* Left-bundle branch block or significant ST-T wave changes on the baseline ECG without a perfusion stress test, demonstrating no reversible ischemia within the 3 months before study entry
* Stopping during the treadmill exercise stress test because of chest pain, shortness of breath, hip or knee arthritis. These individuals will be interviewed by the principal investigator and will be excluded only if it is determined that their walking performance (based in part on the treadmill test) is limited by a comorbidity other than leg ischemia.
* Unable to walk at least 50 feet without stopping during the 6-minute walk test
* Stopping during the 6-minute walk test for symptoms other than ischemic leg symptoms
* Mini-Mental Status Examination (MMSE) score of less than 23 or psychiatric illness
* Failure to complete a study run-in period
* Parkinson's disease
* Requires oxygen with exertion.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2008-06; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
6-minute walk test at 6 month follow-up | Measured at baseline and Month 6 follow-up

SECONDARY OUTCOMES:
Treadmill walking performance | Measured at baseline and Month 6 follow-up
Health-related quality of life measures | Measured at baseline, Month 6, and Month 12 follow-up
Physical activity levels | Measured at baseline, Month 6, and Month 12 follow-up
6-minute walk test at Month 12 follow-up | Measured at Month 12 follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mary M. McDermott, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Derived] Kosmac K, Gonzalez-Freire M, McDermott MM, White SH, Walton RG, Sufit RL, Tian L, Li L, Kibbe MR, Criqui MH, Guralnik JM, S Polonsky T, Leeuwenburgh C, Ferrucci L, Peterson CA. Correlations of Calf Muscle Macrophage Content With Muscle Properties and Walking Performance in Peripheral Artery Disease. J Am Heart Assoc. 2020 May 18;9(10):e015929. doi: 10.1161/JAHA.118.015929. Epub 2020 May 9. PMID 32390569
- [Derived] McDermott MM, Guralnik JM, Criqui MH, Ferrucci L, Liu K, Spring B, Tian L, Domanchuk K, Kibbe M, Zhao L, Lloyd Jones D, Liao Y, Gao Y, Rejeski WJ. Unsupervised exercise and mobility loss in peripheral artery disease: a randomized controlled trial. J Am Heart Assoc. 2015 May 20;4(5):e001659. doi: 10.1161/JAHA.114.001659. PMID 25994445
- [Derived] McDermott MM, Guralnik JM, Criqui MH, Ferrucci L, Zhao L, Liu K, Domanchuk K, Spring B, Tian L, Kibbe M, Liao Y, Lloyd Jones D, Rejeski WJ. Home-based walking exercise in peripheral artery disease: 12-month follow-up of the GOALS randomized trial. J Am Heart Assoc. 2014 May 21;3(3):e000711. doi: 10.1161/JAHA.113.000711. PMID 24850615
- [Derived] Rejeski WJ, Spring B, Domanchuk K, Tao H, Tian L, Zhao L, McDermott MM. A group-mediated, home-based physical activity intervention for patients with peripheral artery disease: effects on social and psychological function. J Transl Med. 2014 Jan 28;12:29. doi: 10.1186/1479-5876-12-29. PMID 24467875
- [Derived] McDermott MM, Liu K, Guralnik JM, Criqui MH, Spring B, Tian L, Domanchuk K, Ferrucci L, Lloyd-Jones D, Kibbe M, Tao H, Zhao L, Liao Y, Rejeski WJ. Home-based walking exercise intervention in peripheral artery disease: a randomized clinical trial. JAMA. 2013 Jul 3;310(1):57-65. doi: 10.1001/jama.2013.7231. PMID 23821089